CLINICAL TRIAL: NCT01219179
Title: The Use of Enteral Sterile Water Feeds for the Treatment of Hypernatremia in Extremely Low Birth Weight Infants
Brief Title: Use of Sterile Water Feeds for Treatment of Hypernatremia in Extremely Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Amy Bieda, Student, Case Western Reserve University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-10-22
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Extremely Low Birth Weight Infants; Hypernatremia
Keywords: Extremely Low Birth Weight Infants; Hypernatremia; Enteral Sterile Water Feeds
MeSH Terms: conditions — Hypernatremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sterile water (Experimental): Intervention group received sterile water if their sodium value was greater or equal to 150 mEq/liter
  Interventions: Other: Sterile water feedings

INTERVENTIONS:
Other: Sterile water feedings — Control group- no intervention
  Prophylactic group will receive sterile water feeds starting at 24 hours of life if/or when their serum sodium value is ≥ 145 mEq/L. The volume of sterile water is 10mls/Kg/day based on birth weight, given via continuous infusion feed.
  The feeding will be stopped when the serum sodium value is ≤ 140 mEq/L.
  The hypernatremia group will receive sterile water feeds when their serum sodium value is ≥ 150 meq/L. The volume of sterile water is 10 mls/Kg/day based on birth weight,given via continuous infusion feed. The feeding will be stopped when the serum sodium value is ≤ 140 mEq/L.

SUMMARY:
The improved survival rate of extremely low birth weight(ELBW)infants has resulted in new fluid and electrolyte problems that have not been encountered previously,in particular electrolyte imbalance. ELBW infants are especially vulnerable to hypernatremia(serum sodium value >150 mEq/L). Hypernatremia may be due to rapid dehydration or excessive administration of intravenous fluids(IV)that contain sodium. The current treatment modality for hypernatremia is to increase IV fluids above daily requirements.Enteral sterile water feeds(ESWF)are theorized as an endogenous source of fluids that may decrease elevated electrolytes such as sodium and potassium in premature infants. By giving ESWF to decrease elevated electrolytes, there would be less need for large volumes of IVF that contribute to the co-morbidities of prematurity: bronchopulmonary dysplasia (BPD),intraventricular hemorrhage(IVH)and patent ductus arteriosus(PDA).

The purpose of this proposed study is to determine whether enteral sterile water feedings is effective in decreasing the incidence, duration and severity of hypernatremia in ELBW infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than or equal to 1,100 grams birth weight
* Less than or equal to 28 weeks gestational age

Exclusion Criteria:

* * Congenital heart disease, other than a PDA

  * Major congenital anomalies
  * A surgical condition (gastroschisis,omphalocele)
  * Renal disease
  * Hypotension treated with pressor support
  * Reverse end diastolic flow on Doppler study prior to delivery
  * Emergency medication received in the delivery room,except fluid boluses
  * Apgar scores recorded at 10 minutes of life < or up to 5 and/or pH less than 7.0 on the first blood gas upon admission to the NICU

Ages: 24 Hours to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
serum sodium values | Every 12 hours for 7 days
  electrolytes will be measured every 12 hours from admission through the first seven days of life

CONTACTS AND LOCATIONS:
Overall Officials: Donna Dowling, PhD, Study Chair — Case Western Reserve University
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States